CLINICAL TRIAL: NCT02624752
Title: Nutrition Supplementation in Hospitalized Patients (NutriSup Oral)
Brief Title: Oral Nutrition Supplementation in Hospitalized Patients
Acronym: NutriSup Oral
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIG2014F-08B
Record Dates: First submitted 2015-12-04; First posted 2015-12-08 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Malnutrition
Keywords: Oral Nutrition Supplementation
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Patients will be randomized via REDCap (Research Electronic Data Capture), a secure, centralized web-based randomization module to:
  1. Ensure Enlive (enhanced ONS) + standard menu; or
  2. Standard of care (including standard menu and possibly ONS) Patients randomized will receive standard menu or standard menu plus enhanced oral nutritional supplements (ONS). Patients randomized to enhanced ONS, will receive one bottle of ONS Abbott Ensure Enlive (235 mL, 350 calories), or similar product, two times daily for 90 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of care could include liberalized diet consisting of 3 meals and snacks served daily or the standard oral nutrition supplementation (ONS) routinely used in the hospital, as prescribed by the medical team.These routine meals and snacks are the "standard of care."
- Ensure (Experimental): Patients randomized to Enhanced Oral Nutritional Supplementation (ONS) will receive the standard of care hospital menu (3 meals and snacks per day) plus 2 cans of Ensure (or similar product) per day while in hospital and will continue 2 cans per day of Ensure when discharged home until they have been receiving the enhanced ONS for a total of 90 days.
  Interventions: Dietary Supplement: Ensure

INTERVENTIONS:
Dietary Supplement: Ensure — Comparison of enhanced oral nutrition supplementation versus standard of care
  Arms: Ensure

SUMMARY:
The purpose of this pilot study is to determine the effect of 3 months use of enhanced Oral Nutritional Supplement (ONS) on physical function and functional performance in malnourished elderly patients.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine the effect of 3 months use of enhanced Oral Nutritional Supplementation (ONS) on muscle accretion and functional performance in malnourished elderly patients. The objectives of this study are to determine feasibility of recruitment, adherence to intervention and retention of the sample, as well as the capacity of subjects to complete functional and muscle mass measures for a planned multi-centre Randomized Controlled Trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* admitted to a general medical ward and recruited within 48 hours
* over the age of 65 years
* malnourished (subjective global assessment categories B or C patients)

Exclusion Criteria:

* have an allergy or intolerance to any component of the oral supplement
* are designated palliative care
* are currently suffering from refeeding syndrome
* have a pre-existing medical condition that prevents oral intake of full fluids,
* have an expected length of stay of less than 48 hours from the time of assessment
* have suspected ischemic stroke as cause for admission
* reside in a residential care home
* are unable to walk prior to current illness.
* are pregnant/breastfeeding
* have a current diagnosis of diabetic ketoacidosis or hyperglycemic hyperosmolar syndrome

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Hospital Readmission Rate | 90 days
  The number of participants who are re-admitted to hospital within 90 days of randomization. This healthcare utilization outcome will be used to determine the cost-benefit of enhanced Oral Nutritional Supplementation.

SECONDARY OUTCOMES:
Successful recruitment | 1 year
  We will view this pilot study as demonstrating feasibility of recruitment if we are able to recruit 60 patients over twelve months (approximately 5 patients per month for the overall study).
Adherence to treatment | 90 days
  Adherence to the study treatments will be defined as ≥85% of patients were given the allocated intervention. Preliminary estimates of non-administration of the trial intervention are needed, along with strategies that maximize exposure to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Rahman, MD, FRCPC, Principal Investigator — St.Joseph's Health Care, London ON
Locations (1):
- LHSC-University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No